CLINICAL TRIAL: NCT01606956
Title: The Comparison of Two Different Methods of Partial Inflation of Cuff for Facile Insertion of Laryngeal Mask Airway in Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 1-2012-0012
Record Dates: First submitted 2012-05-22; First posted 2012-05-28 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: General Anesthesia

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- resting volume group (Experimental)
  Interventions: Procedure: The cuff inflation by the resting volume
- half the maximum volume group (Active Comparator)
  Interventions: Procedure: The cuff inflation by half the maximum volume

INTERVENTIONS:
Procedure: The cuff inflation by the resting volume — 80 patients are randomly allocated into two groups : resting volume group (n=40), half the maximum volume group (n=40). In the resting volume group, the pilot balloon valve is connected to syringe without piston for keeping the valve open to the atmosphere and allowing the pressure within the cuff of LMA to equalize with atmospheric pressure. In the half the maximum volume group, the cuff of LMA is completely emptied and then the cuff is filled with the half the maximum volume.
  Arms: resting volume group
Procedure: The cuff inflation by half the maximum volume — 80 patients are randomly allocated into two groups : resting volume group (n=40), half the maximum volume group (n=40). In the resting volume group, the pilot balloon valve is connected to syringe without piston for keeping the valve open to the atmosphere and allowing the pressure within the cuff of LMA to equalize with atmospheric pressure. In the half the maximum volume group, the cuff of LMA is completely emptied and then the cuff is filled with the half the maximum volume.
  Arms: half the maximum volume group

SUMMARY:
Partial cuff inflation before insertion is generally used for laryngeal mask airway insertion in adult patients. However, it is not proven how much the cuff should be inflated. The aim of this study is to compare efficacy between the method using the resting volume and the method using half the maximum volume for partial cuff inflation.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (20-70 years of age) scheduled for elective surgery undergoing general anesthesia using LMA-classic size 3-5

Exclusion Criteria:

* patients with an abnormal airway,
* patients with reactive airway disease,
* patients with gastroesophageal reflux disease,
* patients with chronic respiratory disease,
* or a history of an upper respiratory tract infection

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The intra-cuff pressure | approximately 5 to 10 minutes after insertion of LMA.
  After insertion of LMA, we confirm adequate ventilation. And then we measure intra-cuff pressure using cuff pressure manometer.

SECONDARY OUTCOMES:
leak volume | approximately 5 to 10 minutes after insertion of LMA.
  After confirming adequate ventilation, tidal volumes are measured using spirometer sensor attached anesthesia machine. Five corresponding inspiratory and expiratory tidal volumes are recorded and the difference between these is calculated as the leak volume.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Al-Shaikh B, George William M, Van Zundert AA. Using atmospheric pressure to inflate the cuff of the Portex Laryngeal Mask. Anaesthesia. 2005 Mar;60(3):296-7. doi: 10.1111/j.1365-2044.2005.04135.x. No abstract available. PMID 15710025
- [Derived] Kim MS, Lee JR, Shin YS, Chung JW, Lee KH, Ahn KR. Comparison of 2 cuff inflation methods of laryngeal mask airway Classic for safe use without cuff manometer in adults. Am J Emerg Med. 2014 Mar;32(3):237-42. doi: 10.1016/j.ajem.2013.11.029. Epub 2013 Nov 21. PMID 24360025